CLINICAL TRIAL: NCT06975774
Title: Randomized, Double-blind, Double-mal Injection, Control Study of Phase II Clinical Dose Calibration of BCG Pure Protein Derivative (BCG-PPD)
Brief Title: Phase II Clinical Clical of the Pure Protein Derivatives of BCG
Acronym: BCG-PPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Shenzhen Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2021-PPD01
Record Dates: First submitted 2024-12-06; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-12

CONDITIONS: Tuberculosis
Keywords: diagnosis of tuberculosis; epidemiological investigation of tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCG-PPD under test Is applied to the left arm, while the marketed BCG-PPD Is applied to the right (Experimental): Thirty subjects were randomized, double-blinded to perform a homogeneous double-arm BCG-PPD skin test
  Interventions: Drug: Purified Protein Derivative of BCG（BCG-PPD）
- BCG-PPD under test Is applied to the right arm, while the marketed BCG-PPD Is applied to the left (Experimental): Thirty subjects were randomized, double-blinded to perform a homogeneous double-arm BCG-PPD skin test
  Interventions: Drug: Purified Protein Derivative of BCG（BCG-PPD）

INTERVENTIONS:
Drug: Purified Protein Derivative of BCG（BCG-PPD） — Thirty subjects were randomized, double-blinded to perform a homogeneous double-arm BCG-PPD skin test.

SUMMARY:
This phase II clinical trial used randomized, double-blind, double-arm intradermal injection, and the same marketed products, selected 30 pulmonary tuberculosis patients aged 18-65 years who met the inclusion criteria and did not meet the exclusion criteria, and conducted the double-arm skin test using BCG-PPD and marketed BCG-PPD controls.

During the screening period, the subjects underwent evidence collection of confirmed tuberculosis, physical examination, vital signs, blood routine, urine routine, blood biochemistry, electrocardiogram, chest CT, HIV antibody test, and blood pregnancy examination of women of childbearing age; Vital signs examination before the skin test, The injection site was photographed 0min after the skin test, Vital signs were performed 30min after the skin test; Vital signs were examined, pictures of the injection site was taken, and the injection site reaction was measured; Observe the skin test response, Record the redness, hardening longitudinal diameter and transverse diameter and other related reactions; All adverse events within 72h after the skin test were recorded and safety evaluated.

DETAILED DESCRIPTION:
Prior to the commencement of the study, the Investigator/his authorized officer will contact the subject and/or guardian to enroll the candidate subjects and invite them to participate in the study.Subjects who are eligible for screening receive the drug number in the order they arrive at the random number allocation room.During the screening period, tuberculosis diagnosis evidence collection, physical examination, vital signs, blood routine, urine routine test, blood biochemistry, electrocardiogram, chest CT, HIV antibody test and blood pregnancy examination of women of childbearing age were conducted; after screening, study number (drug number) was assigned, and double arm BCG-PPD skin test with 0.1ml injection. Vital signs should be taken before skin test, injection site photographed 0min and 30min after skin test; vital signs examined, injection site photographed and measured 48-72h after skin test; observe skin test reaction, record red, hard vertical diameter and transverse diameter and other related reactions of skin test; record all adverse events within 72h after skin test and perform safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* The subject shall be judged as a confirmed tuberculosis patient by a clinician according to Section 5.3.1-5.3.6 of the Health Industry Standards of the People's Republic of China (WS288-2017) (Annex I).(The sampling time can be accepted for the laboratory examination is the examination results of the hospital within 30 days before the skin test);
* Age 18~65, male or female;
* I agree to participate in this trial and sign the informed consent form;
* I am able to follow the follow-up requirements of the clinical trial protocol for follow-up

Exclusion Criteria:

* People suffering from acute infectious diseases (such as measles, whooping cough, influenza, pneumonia, etc.), acute ocular conjunctivitis, acute otitis media, extensive skin diseases and allergic constitution;
* Having serious diseases not considered suitable for enrollment by the investigator, such as: advanced tumor, acute onset of chronic obstructive pulmonary disease, acute or progressive liver disease or kidney disease, congestive heart failure, etc.;
* Those treated with immunosuppressants or immune enhancer, or those receiving glucocorticoids, immunoglobulin preparations other than the gastrointestinal tract, or blood products or plasma extracts within 1 month;
* Those who are participating in other new drug clinical trials or have participated in any other new drug clinical trials within 3 months before the clinical trial;
* Women during pregnancy or lactation;
* Patients with mental illness onset period;
* PPD or similar products within 3 months;
* The investigator considered poor compliance, past history, physical examination or laboratory findings.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Injection-site reaction endpoint | Within 24 hours and 48 hours to 72 hours after the skin test
  Evaluate the occurrence of positive reactions，like the transverse and longitudinal diameter of skin redness, induration, and strong positive reactions in 24 hours necrosis, and lymphangitis between 24 hours and 72 hours after the skin test
Safety endpoint | Within 72 hours after the skin test
  The incidence of all adverse events (AES) within 72 hours after drug injection in the subjects;

CONTACTS AND LOCATIONS:
Overall Officials: Lu Shuihua, Bachelor, Principal Investigator — Shenzhen Third People's Hospital
Locations (1):
- The Third People's Hospital Of Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No